CLINICAL TRIAL: NCT02242331
Title: Risk of Morning Hypertension
Brief Title: Post-marketing Study to Supplement Data on Safety, Tolerability and Efficacy of Micardis® With Special Emphasis on the Control of Blood Pressure
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.386
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- essential hypertension patients
  Interventions: Drug: Micardis®

INTERVENTIONS:
Drug: Micardis®

SUMMARY:
This post-marketing surveillance study is designed to supplement under conditions of normal clinical practice data on safety, tolerability and efficacy of Micardis® collected in clinical studies with special emphasis on the control of blood pressure in the morning before intake of the next antihypertensive drug

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension
* At least 18 years of age

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of essential hypertension recruited at general practitioners and specialists in internal medicine in non-hospital practice
Sampling Method: Non-Probability Sample
Enrollment: 19805 (Actual)
Dates: Start 2001-06; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood pressure | Baseline, after 3 months
  with special emphasis on the morning blood pressure, before intake of the next antihypertensive treatment
Number of patients with adverse events | up to 3 months
Changes from baseline in pulse rate | Baseline, after 3 months

SECONDARY OUTCOMES:
Assessment of efficacy by investigator on 5- point scale | after 3 months
Assessment of tolerability by investigator on a 5-point scale | after 3 months